CLINICAL TRIAL: NCT01922999
Title: A Randomized, Prospective, Double Blind, Placebo-Controlled Trial of Two Different Doses of Oral Melatonin Supplements in Chronic Kidney Disease (CKD)-Associated Sleep Disorders
Brief Title: Different Doses of Oral Melatonin Supplements in Chronic Kidney Disease (CKD)-Associated Sleep Disorders
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast Renal Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Melatonin
Record Dates: First submitted 2013-08-07; First posted 2013-08-14 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: End Stage Renal Disease; Chronic Kidney Disease; Sleep Disorder
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Sleep Wake Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo controlled (Active Comparator): comparison of placebo controlled to 1mg melatonin or 3mg melatonin
  Interventions: Drug: Melatonin
- Melatonin (Active Comparator): comparison of melatonin 1mg or melatonin 3mg
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — patients will receive placebo, 1mg melatonin or 3mg melatonin

SUMMARY:
The study will evaluate the safety and efficacy of melatonin supplementation in CKD and ESRD patients with sleep disorders to reduce sleep latency times, the number of apnea/hypopneic episodes, and prolong duration in rapid eye movement (REM) sleep in CKD and ESRD patients with sleep disordered breathing.

DETAILED DESCRIPTION:
The study will look at the safety and efficacy of melatonin supplementation given to patients with chronic kidney disease and end stage renal disease who have sleep disorders to reduce sleep latency times, the number of apnea/hypopneic episodes, and prolong duration in rapid eye movement (REM) sleep in CKD and ESRD patients with sleep disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age > 18 and <85 years of age
2. Patients with CKD or ESRD with eGFR < 30 mls/min
3. If receiving hemodialysis, patients must be on treatment > 3 months
4. Normal healthy controls must be without a known history of CKD and be willing to have formal PSG test and plasma melatonin measurements

Exclusion Criteria:

1. Patients receiving outpatient hemodialysis for < 3 months
2. Patients with estimated GFR by Cockcroft Gault > 30 mls/min
3. Patients receiving beta blocker therapy within one month of randomization
4. Patients receiving Nifedipine therapy within one month randomization
5. Patients on peritoneal dialysis
6. Patient with chronic home oxygen supplementation
7. Patients receiving chronic home CPAP therapy
8. Patients actively receiving outpatient sleep medications
9. Patients with diabetic gastroparesis unresponsive to medication
10. Patients with known pregnancy or unwilling to use contraception during the course of the study
11. Patients with a functioning renal allograft
12. Patient currently receiving long-term immunosuppressive therapy. Patients receiving low dose prednisone (10mg or less per day) will not be excluded from this trial
13. Unable to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2012-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | Compare sleep duration at the end of 60 days
  Patients taking melatonin supplement, 1mg or 3mg daily, compared to placebo controlled group will be compared to see who group achieved a 25% reduction in sleep latency or 25% increase in total sleep time at the end of 60 days. Using the Pittsburg Sleep Quality Index (PSQI) questionnaire as the index to measure quality of sleep and sleep patterns. Study will also use Polysomnography testing that will record duration of sleep patterns.

CONTACTS AND LOCATIONS:
Overall Officials: James A Tumlin, MD, Principal Investigator — Southeast Renal Research Institute
Locations (1):
- Southeast Renal Research Institute, Chattanooga, Tennessee, United States